CLINICAL TRIAL: NCT06871540
Title: Evaluation of the Effect of Streptococcus Salivarius K12 Probiotic in the Treatment of Periodontitis: a Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Effect of Streptococcus Salivarius K12 Probiotic in the Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AYŞENUR ŞAHİN (Other)
Responsible Party: Sponsor-Investigator, AYŞENUR ŞAHİN, Research assistant, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: INU-DHF-AS-01
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis Stage III; Probiotic
Keywords: Microbiology, Periodontitis, Probiotics, Cytokines
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Grubu (Active Comparator)
  Interventions: Other: Probiotic Agent; Other: Non-Surgical Intervention
- Control (Other)
  Interventions: Other: Non-Surgical Intervention

INTERVENTIONS:
Other: Probiotic Agent — Patients in the test group were instructed to take one tablet immediately after tooth brushing (before bedtime) once daily for 30 consecutive days. Probiotic was administered in tablets containing 1x109 cfu/g S. salivarius K12.
  Arms: Test Grubu
Other: Non-Surgical Intervention — Patients in the control group received non-surgical periodontal treatment only.

SUMMARY:
Aims: The use of oral probiotics as an adjunct to the treatment of periodontal diseases is known to be beneficial in antagonizing pathogenic microflora and regulating the host immune response. The aim of this clinical study was to evaluate the clinical, microbiologic and biochemical effect of Streptococcus salivarius (S. salivarius) K12 probiotic tablet as an adjunct to scaling and root planing (SRP) treatment in stage 3 periodontitis patients.

Methods: The study included 30 systemically healthy stage 3 periodontitis patients. After non-surgical periodontal treatment, participants were randomly assigned to the test (SRP+Probiotic, n=15) or control (SRP, n=15) group. Patients in the test group used probiotic tablets once daily for 30 days. Clinical (Plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing depth (PD), clinical attachment level (CAL)), microbiological (Porphyromonas gingivalis, Treponema denticola, Tannerella forsythia, Prevotella intermedia, Aggregatibacter actinomycetemcomitans, Fusobacterium nucleatum) and biochemical (IL-6, IL-8, IL-10) measurements were performed at baseline (before SRP), 30. and 90th days. Data were analyzed statistically.

Keywords: Microbiology, Periodontitis, Probiotics, Cytokines

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-60 years,
* No systemic disease,
* No periodontal treatment in the last 6 months,
* No antibiotic therapy in the last 6 months,
* Diagnosed with stage 3 periodontitis according to the 2017 periodontal disease classification

Exclusion Criteria:

* Periodontal treatment within sixteen months,
* Smoking,
* Patients with systemic health problems such as diabetes, rheumatoid arthritis, neurological diseases, lung and kidney diseases,
* Pregnancy or lactation,
* Acute oral lesions or necrotizing ulcerative periodontitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in Porphyromonas gingivalis at 3 months | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- İnönü Üniversitesi Diş Hekimliği Fakültesi, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haffajee AD, Cugini MA, Dibart S, Smith C, Kent RL Jr, Socransky SS. Clinical and microbiological features of subjects with adult periodontitis who responded poorly to scaling and root planing. J Clin Periodontol. 1997 Oct;24(10):767-76. doi: 10.1111/j.1600-051x.1997.tb00195.x. PMID 9350562
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Background] Servin AL, Coconnier MH. Adhesion of probiotic strains to the intestinal mucosa and interaction with pathogens. Best Pract Res Clin Gastroenterol. 2003 Oct;17(5):741-54. doi: 10.1016/s1521-6918(03)00052-0. PMID 14507585
- [Background] Morales A, Carvajal P, Silva N, Hernandez M, Godoy C, Rodriguez G, Cabello R, Garcia-Sesnich J, Hoare A, Diaz PI, Gamonal J. Clinical Effects of Lactobacillus rhamnosus in Non-Surgical Treatment of Chronic Periodontitis: A Randomized Placebo-Controlled Trial With 1-Year Follow-Up. J Periodontol. 2016 Aug;87(8):944-52. doi: 10.1902/jop.2016.150665. Epub 2016 Mar 4. PMID 26944407
- [Background] Darveau RP, Hajishengallis G, Curtis MA. Porphyromonas gingivalis as a potential community activist for disease. J Dent Res. 2012 Sep;91(9):816-20. doi: 10.1177/0022034512453589. Epub 2012 Jul 6. PMID 22772362
- [Background] Stamatova I, Meurman JH. Probiotics and periodontal disease. Periodontol 2000. 2009;51:141-51. doi: 10.1111/j.1600-0757.2009.00305.x. No abstract available. PMID 19878473
- [Background] Alanzi A, Honkala S, Honkala E, Varghese A, Tolvanen M, Soderling E. Effect of Lactobacillus rhamnosus and Bifidobacterium lactis on gingival health, dental plaque, and periodontopathogens in adolescents: a randomised placebo-controlled clinical trial. Benef Microbes. 2018 Jun 15;9(4):593-602. doi: 10.3920/BM2017.0139. Epub 2018 Apr 10. PMID 29633646
- [Background] Twetman S, Derawi B, Keller M, Ekstrand K, Yucel-Lindberg T, Stecksen-Blicks C. Short-term effect of chewing gums containing probiotic Lactobacillus reuteri on the levels of inflammatory mediators in gingival crevicular fluid. Acta Odontol Scand. 2009;67(1):19-24. doi: 10.1080/00016350802516170. PMID 18985460
- [Background] Rossi V, Romagna R, Angst PDM, Gomes SC. Gingival crevicular fluid response to protocols of non-surgical periodontal therapy: A longitudinal evaluation. Indian J Dent Res. 2019 Sep-Oct;30(5):736-741. doi: 10.4103/ijdr.IJDR_148_16. PMID 31854365
- [Background] Kowashi Y, Jaccard F, Cimasoni G. Sulcular polymorphonuclear leucocytes and gingival exudate during experimental gingivitis in man. J Periodontal Res. 1980 Mar;15(2):151-8. doi: 10.1111/j.1600-0765.1980.tb00269.x. No abstract available. PMID 6445977
- [Background] Ince G, Gursoy H, Ipci SD, Cakar G, Emekli-Alturfan E, Yilmaz S. Clinical and Biochemical Evaluation of Lozenges Containing Lactobacillus reuteri as an Adjunct to Non-Surgical Periodontal Therapy in Chronic Periodontitis. J Periodontol. 2015 Jun;86(6):746-54. doi: 10.1902/jop.2015.140612. Epub 2015 Mar 5. PMID 25741580
- [Background] Laleman I, Yilmaz E, Ozcelik O, Haytac C, Pauwels M, Herrero ER, Slomka V, Quirynen M, Alkaya B, Teughels W. The effect of a streptococci containing probiotic in periodontal therapy: a randomized controlled trial. J Clin Periodontol. 2015 Nov;42(11):1032-41. doi: 10.1111/jcpe.12464. Epub 2015 Nov 29. PMID 26427036
- [Background] Tekce M, Ince G, Gursoy H, Dirikan Ipci S, Cakar G, Kadir T, Yilmaz S. Clinical and microbiological effects of probiotic lozenges in the treatment of chronic periodontitis: a 1-year follow-up study. J Clin Periodontol. 2015 Apr;42(4):363-72. doi: 10.1111/jcpe.12387. Epub 2015 Apr 10. PMID 25728888
- [Background] Teughels W, Durukan A, Ozcelik O, Pauwels M, Quirynen M, Haytac MC. Clinical and microbiological effects of Lactobacillus reuteri probiotics in the treatment of chronic periodontitis: a randomized placebo-controlled study. J Clin Periodontol. 2013 Nov;40(11):1025-35. doi: 10.1111/jcpe.12155. Epub 2013 Sep 15. PMID 24164569
- [Background] Vivekananda MR, Vandana KL, Bhat KG. Effect of the probiotic Lactobacilli reuteri (Prodentis) in the management of periodontal disease: a preliminary randomized clinical trial. J Oral Microbiol. 2010 Nov 2;2. doi: 10.3402/jom.v2i0.5344. PMID 21523225
- [Background] Krasse P, Carlsson B, Dahl C, Paulsson A, Nilsson A, Sinkiewicz G. Decreased gum bleeding and reduced gingivitis by the probiotic Lactobacillus reuteri. Swed Dent J. 2006;30(2):55-60. PMID 16878680
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] MacDonald KW, Chanyi RM, Macklaim JM, Cadieux PA, Reid G, Burton JP. Streptococcus salivarius inhibits immune activation by periodontal disease pathogens. BMC Oral Health. 2021 May 7;21(1):245. doi: 10.1186/s12903-021-01606-z. PMID 33962608
- [Background] Burton JP, Wescombe PA, Cadieux PA, Tagg JR. Beneficial microbes for the oral cavity: time to harness the oral streptococci? Benef Microbes. 2011 Jun;2(2):93-101. doi: 10.3920/BM2011.0002. PMID 21840808
- [Background] Meurman JH, Stamatova I. Probiotics: contributions to oral health. Oral Dis. 2007 Sep;13(5):443-51. doi: 10.1111/j.1601-0825.2007.01386.x. PMID 17714346
- [Background] Shah MP, Gujjari SK, Chandrasekhar VS. Evaluation of the effect of probiotic (inersan(R)) alone, combination of probiotic with doxycycline and doxycycline alone on aggressive periodontitis - a clinical and microbiological study. J Clin Diagn Res. 2013 Mar;7(3):595-600. doi: 10.7860/JCDR/2013/5225.2834. Epub 2013 Mar 1. PMID 23634432
- [Background] Iniesta M, Herrera D, Montero E, Zurbriggen M, Matos AR, Marin MJ, Sanchez-Beltran MC, Llama-Palacio A, Sanz M. Probiotic effects of orally administered Lactobacillus reuteri-containing tablets on the subgingival and salivary microbiota in patients with gingivitis. A randomized clinical trial. J Clin Periodontol. 2012 Aug;39(8):736-44. doi: 10.1111/j.1600-051X.2012.01914.x. Epub 2012 Jun 13. PMID 22694350
- [Background] Staab B, Eick S, Knofler G, Jentsch H. The influence of a probiotic milk drink on the development of gingivitis: a pilot study. J Clin Periodontol. 2009 Oct;36(10):850-6. doi: 10.1111/j.1600-051X.2009.01459.x. Epub 2009 Aug 12. PMID 19682173
- [Background] Maassen CB, van Holten-Neelen C, Balk F, den Bak-Glashouwer MJ, Leer RJ, Laman JD, Boersma WJ, Claassen E. Strain-dependent induction of cytokine profiles in the gut by orally administered Lactobacillus strains. Vaccine. 2000 May 22;18(23):2613-23. doi: 10.1016/s0264-410x(99)00378-3. PMID 10775795
- [Background] Salminen S, Benno Y, de Vos W. Intestinal colonisation, microbiota and future probiotics? Asia Pac J Clin Nutr. 2006;15(4):558-62. PMID 17077076
- [Background] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Background] Teughels W, Van Essche M, Sliepen I, Quirynen M. Probiotics and oral healthcare. Periodontol 2000. 2008;48:111-47. doi: 10.1111/j.1600-0757.2008.00254.x. No abstract available. PMID 18715361
- [Background] Kapoor A, Malhotra R, Grover V, Grover D. Systemic antibiotic therapy in periodontics. Dent Res J (Isfahan). 2012 Sep;9(5):505-15. doi: 10.4103/1735-3327.104866. PMID 23559912
- [Background] Hanes PJ, Purvis JP. Local anti-infective therapy: pharmacological agents. A systematic review. Ann Periodontol. 2003 Dec;8(1):79-98. doi: 10.1902/annals.2003.8.1.79. PMID 14971250
- [Background] Quirynen M, Teughels W, De Soete M, van Steenberghe D. Topical antiseptics and antibiotics in the initial therapy of chronic adult periodontitis: microbiological aspects. Periodontol 2000. 2002;28:72-90. doi: 10.1034/j.1600-0757.2002.280104.x. No abstract available. PMID 12013349
- [Background] Yen CA, Damoulis PD, Stark PC, Hibberd PL, Singh M, Papas AS. The effect of a selective cyclooxygenase-2 inhibitor (celecoxib) on chronic periodontitis. J Periodontol. 2008 Jan;79(1):104-13. doi: 10.1902/jop.2008.070271. PMID 18166099
- [Background] Okada H, Murakami S. Cytokine expression in periodontal health and disease. Crit Rev Oral Biol Med. 1998;9(3):248-66. doi: 10.1177/10454411980090030101. PMID 9715365
- [Background] Haffajee AD, Socransky SS. Microbial etiological agents of destructive periodontal diseases. Periodontol 2000. 1994 Jun;5:78-111. doi: 10.1111/j.1600-0757.1994.tb00020.x. No abstract available. PMID 9673164
- [Background] Berezow AB, Darveau RP. Microbial shift and periodontitis. Periodontol 2000. 2011 Feb;55(1):36-47. doi: 10.1111/j.1600-0757.2010.00350.x. No abstract available. PMID 21134227
- [Background] Slots J. Periodontitis: facts, fallacies and the future. Periodontol 2000. 2017 Oct;75(1):7-23. doi: 10.1111/prd.12221. PMID 28758294